CLINICAL TRIAL: NCT05958914
Title: Evaluation of Neuropeptide Expression During the Ovarian Cycle and in Patients With PCOS: Pilot Study
Brief Title: Neuropeptide Expression During the Ovarian Cycle and in Patients With PCOS
Acronym: PCO-NP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Sandro Gerli, Associate Professor of Obstetrics and Gynecology, University Of Perugia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 27139
Record Dates: First submitted 2023-06-12; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: PCOS
Keywords: PCOS; neuropeptides; enkephalins; SP; CGRP; VIP

STUDY DESIGN:
Intervention Model Description: The study involves an enrollment of 45 total patients, referred to the Medically assisted reproduction Center, divided into 3 groups, of 15 patients each: Group 1 (control) women with regular ovarian cycle; Group 2- non-PCOS women undergoing ovarian stimulation and ICSI treatment; Group 3- women with PCOS undergoing ovarian stimulation and ICSI treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): women with regular ovarian cycle. Patients, as per normal clinical practice, will undergo three blood draws in the follicular, ovulatory and luteal phases.
  Biological samples will be analyzed for the concentration of neuropeptides (enkephalins, CGRP, SP and VIP)
  Interventions: Diagnostic Test: Dosage of ematic CGRP; Diagnostic Test: Dosage of ematic SP; Diagnostic Test: Dosage of ematic enkephalins; Diagnostic Test: Dosage of ematic VIP
- Arm 2 (Experimental): non-PCOS women undergoing ovarian stimulation and ICSI treatment. Patients will undergo ovarian stimulation treatment with gonadotropins and egg retrieval. As part of this process, as per clinical practice, blood and follicular fluid sampling will be performed.
  Biological samples will be analyzed for the concentration of neuropeptides (enkephalins, CGRP, SP and VIP)
  Interventions: Diagnostic Test: Dosage of ematic CGRP; Diagnostic Test: Dosage of ematic SP; Diagnostic Test: Dosage of ematic enkephalins; Diagnostic Test: Dosage of ematic VIP; Diagnostic Test: Dosage of CGRP in follicolar fluid; Diagnostic Test: Dosage of SP in follicolar fluid; Diagnostic Test: Dosage of enkephalins in follicolar fluid; Diagnostic Test: Dosage of VIP in follicolar fluid
- Arm 3 (Experimental): PCOS women undergoing ovarian stimulation and ICSI treatment. Patients will undergo ovarian stimulation treatment with gonadotropins and egg retrieval. As part of this process, as per clinical practice, blood and follicular fluid sampling will be performed.
  Biological samples will be analyzed for the concentration of neuropeptides (enkephalins, CGRP, SP and VIP)
  Interventions: Diagnostic Test: Dosage of ematic CGRP; Diagnostic Test: Dosage of ematic SP; Diagnostic Test: Dosage of ematic enkephalins; Diagnostic Test: Dosage of ematic VIP; Diagnostic Test: Dosage of CGRP in follicolar fluid; Diagnostic Test: Dosage of SP in follicolar fluid; Diagnostic Test: Dosage of enkephalins in follicolar fluid; Diagnostic Test: Dosage of VIP in follicolar fluid

INTERVENTIONS:
Diagnostic Test: Dosage of ematic CGRP — Immunoassay kit for the evaluation of CGRP in blood
Diagnostic Test: Dosage of ematic SP — Immunoassay kit for the evaluation of SP in blood
Diagnostic Test: Dosage of ematic enkephalins — Immunoassay kit for the evaluation of enkephalins in blood
Diagnostic Test: Dosage of ematic VIP — Immunoassay kit for the evaluation of VIP in blood
Diagnostic Test: Dosage of CGRP in follicolar fluid — Immunoassay kit for the evaluation of CGRP in follicolar fluid
  Arms: Arm 2; Arm 3
Diagnostic Test: Dosage of SP in follicolar fluid — Immunoassay kit for the evaluation of SP in follicolar fluid
  Arms: Arm 2; Arm 3
Diagnostic Test: Dosage of enkephalins in follicolar fluid — Immunoassay kit for the evaluation of enkephalins in follicolar fluid
  Arms: Arm 2; Arm 3
Diagnostic Test: Dosage of VIP in follicolar fluid — Immunoassay kit for the evaluation of VIP in follicolar fluid
  Arms: Arm 2; Arm 3

SUMMARY:
The goal of this clinical trial is to characterize PCOS in terms of neuropeptide expression and to make the comparison between women with and without PCOS by going to analyze venous blood samples taken during the three phases of the ovarian cycle and follicular fluid, taken during the ovulatory phase as part of the oocyte pick-up. Specifically, the expression of neuropeptides such as CGRP, SP, VIP and enkephalins in the three phases of the ovarian cycle (follicular phase, ovulatory phase and luteal phase) will be evluated in three groups of women afferent to the medically assisted reproduction centre. In particular, Group 1 (control) will include women with regular ovarian cycle; Group 2 will include non-PCOS women undergoing ovarian stimulation and ICSI treatment; finally Group 3 will include women with PCOS undergoing ovarian stimulation and ICSI treatment.

The main question[s] it aims to answer are:

* Is there a fluctuation in blood neuropeptides concentrations of women with normal ovarian cycles during the three phases of the ovarian cycle?
* Do PCOS women has altered levels of blood and follicolar fluid concentration of neuropepides with respect to non-PCOS individuals?
* Is blood and follicolar fluid concentration of neuropeptide modulated by protocols of ovarian stimulation?

Participants of Group 1 will follow the ovarian monitoring protocol, during which blood samples will be taken at the three phases of the ovarian cycle.

Participants of Group 2 and 3 will undergo ovarian stimulation and ICSI treatment, followed by blood and follicular fluid sampling at the specified cycle phases.

Researchers will compare the control Group 1 with Group 2 and 3 to see if there is a significative difference in the concentration of blood neuropeptides between the three groups at the same phase of the ovarian cycle.

Moreover, they will evaluate if there is there significant different concentration of neuropeptides in follicolar fluid between group 2 and 3 during the ovulatory phase.

DETAILED DESCRIPTION:
This project aims to investigate the neurosensory mechanisms underlying one of the most common disorders related to folliculogenesis, such as PCOS. The study aims to characterize PCOS in terms of neuropeptide expression and to make the comparison between women with and without PCOS, by going to analyze venous blood samples taken during the three phases of the ovarian cycle and follicular fluid, taken during the ovulatory phase as part of the oocyte pick-up. Specifically, the expression of neuropeptides such as CGRP, SP, VIP and enkephalins in the three phases of the ovarian cycle (follicular phase, ovulatory phase and luteal phase) in the three groups of women considered will be evaluated.

Study design:

The study will enroll 45 total patients, referred to the PMA Center, divided into 3 groups of 15 patients each: Group 1 (control) women with regular ovarian cycle; Group 2- non-PCOS women undergoing ovarian stimulation and ICSI treatment; Group 3- women with PCOS undergoing ovarian stimulation and ICSI treatment.

The study will have a total duration of 24 months divided as follows:

* Pre-phase monitoring and enrollment of subjects (20 months).

  * Group 1 will follow the ovarian monitoring protocol, during which blood samples will be taken at the three stages of the ovarian cycle.
  * Group 2 and 3 will undergo ovarian stimulation and ICSI treatment, taken with blood and follicular fluid samples at the specified cycle phases.
* Performance of chemical/biochemical analysis performed at the electrophysiological laboratory of the University of Perugia (2 months).
* Performance of statistical tests and processing of the data obtained (2 months)

Subjects will be given a 4 mL venous blood draw as per regular clinical practice to perform hormone dosing during ovarian cycle monitoring.

No diagnostic tests outside of routine clinical practice are planned, and patients will not be required to travel to the PMA Center for additional visits beyond those required by regular clinical practice.

Subjects and Recruitment Location: 45 patients will be recruited: 15 women with a diagnosis of PCOS and 30 non-PCOS women at the medically assisted reproduction Center of the Perugia Hospital (Head: Prof. S. Gerli).

MATERIALS AND METHODS:

GROUP 1: Patients, as per normal clinical practice, will undergo three blood draws in the follicular, ovulatory and luteal phases.

GROUP 2 and 3: Patients will undergo ovarian stimulation treatment with gonadotropins and egg retrieval. As part of this process, as per clinical practice, blood and follicular fluid sampling will be performed.

Methods Biological Material Collection: During ovarian cycle monitoring, a venous blood sampling will be performed in the morning after at least 10 hours of fasting in patients during the phases described in Table 1. A follicular fluid sample will also be taken during oocyte pick-up (group 2 and 3). Specifically, an aliquot of blood sample, which follicular fluid will be evaluated to assay the level of neuropeptides (CGRP, SP, VIP and enkephalins). The level of CGRP will be measured using an extraction-free enzyme immunoassay kit (Peninsula laboratories LLC, CA, USA) following the manufacturer's protocol. For the quantitative measurement of human substance P, the Human Substance P Enzyme ELISA Assay Kit (ELK1453-96T - Twin Elix srl) will be used. For VIP, the ELISA Kit for Human VIP (ELK1453-96T - Twin Elix srl) will be used, and for the enkephalins assay, the ELISA Kit for Human Enkephalins (ELK5246-96T - Twin Elix srl) will be used. Neuropeptide assays will be conducted at the Physiology Laboratory of the Department of Chemistry, Biology and Biotechnology, University of Perugia, in collaboration with Prof. Fioretti.

Sera will also be analyzed for fasting glucose, triglycerides (TG), total cholesterol (TC), high-density lipoprotein cholesterol (HDL), insulin, dehydroepiandrosterone sulfate (DHEAS), sex hormone-binding globulin (SHBG), progesterone, estradiol, follicle-stimulating hormone (FSH), LH and total testosterone. Serum concentrations of glucose (hexokinase), total cholesterol (CHOD-PAP) and triglycerides (GPO-PAP) will also be measured using standard enzymatic methods (Roche Diagnostics, IN, USA) with a fully automated analyzer (Roche Modular PE, Roche Diagnostics, IN, USA).

ELIGIBILITY:
Inclusion Criteria:

* infertile women
* BMI between 18 and 30 kg/m2,
* basal FSH < 10 IU/L,
* number of antral follicles (2-10 m) per ovary > 10,
* regular uterine cavity assessed by hysterosalpinography, sonohysterography or hysteroscopy, and hematologic and biochemical parameters within normal limits will be included in the study, euthyroid status (with or without treatment)
* In case of women with PCOS, it should be diagnosed according to the Rotterdam criteria (The Rotterdam ESHRE/ASRM-sponsored PCOS consensus workshop group (2004) Revised 2003 consensus on diagnostic criteria and longterm health risks related to polycystic ovary syndrome (PCOS).
* No restrictions regarding the indication of infertility.

Exclusion Criteria:

* presence of ovaries inaccessible to oocyte pick-up,
* presence of sactosalpinx, heterologous fertilization,
* contraindication to pregnancy,
* atypical genital discharge of unspecified cause,
* uncontrolled dystothyroidism, presence of neoplasms,
* severe alteration of liver or kidney function, taking medications that may interfere with the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the normal fluctuation of CGRP during the ovarian cycle in non-PCOS women | 5 days postmenstrual, 14 days postmenstrual, 18 days postmenstrual
  To evaluate the absolute difference of blood concentration of CGRP and the relative difference of its concentration [100 - (CFO*100/CFF) and 100 - (CFL*100/CFO)] in the three phases of the ovarian cycle: follicular phase (FF) (day 5-10 postmenstrual), ovulatory phase (FO) (day 14) and luteal phase (FL) (day 18-23) in women of childbearing age with regular ovarian cycle afferent to the PMA Center (Group 1).
Evaluation of the normal fluctuation of SP during the ovarian cycle in non-PCOS women | 5 days postmenstrual, 14 days postmenstrual, 18 days postmenstrual
  To evaluate the absolute difference of blood concentration of SP and the relative difference of its concentration [100 - (CFO*100/CFF) and 100 - (CFL*100/CFO)] in the three phases of the ovarian cycle: follicular phase (FF) (day 5-10 postmenstrual), ovulatory phase (FO) (day 14) and luteal phase (FL) (day 18-23) in women of childbearing age with regular ovarian cycle afferent to the PMA Center (Group 1).
Evaluation of the normal fluctuation of VIP during the ovarian cycle in non-PCOS women | 5 days postmenstrual, 14 days postmenstrual, 18 days postmenstrual
  To evaluate the absolute difference of blood concentration of VIP and the relative difference of its concentration [100 - (CFO*100/CFF) and 100 - (CFL*100/CFO)] in the three phases of the ovarian cycle: follicular phase (FF) (day 5-10 postmenstrual), ovulatory phase (FO) (day 14) and luteal phase (FL) (day 18-23) in women of childbearing age with regular ovarian cycle afferent to the PMA Center (Group 1).
Evaluation of the normal fluctuation of enkephalins during the ovarian cycle of non PCOS women | 5 days postmenstrual, 14 days postmenstrual, 18 days postmenstrual
  To evaluate the absolute difference of blood concentration of enkephalins and the relative difference of its concentration [100 - (CFO*100/CFF) and 100 - (CFL*100/CFO)] in the three phases of the ovarian cycle: follicular phase (FF) (day 5-10 postmenstrual), ovulatory phase (FO) (day 14) and luteal phase (FL) (day 18-23) in women of childbearing age with regular ovarian cycle afferent to the PMA Center (Group 1).

SECONDARY OUTCOMES:
Evaluation of the fluctuation of CGRP during the ovarian cycle in non-PCOS women undergoing ICSI treatment | 5 days before egg pick-up, day of egg pick up, 10 days after egg pick-up
  Assess the absolute difference of blood concentration of CGRP and the relative difference of its concentration [100 - (CFO*100/CFF) and 100 - (CFL*100/CFO)] in the three phases of the ovarian cycle: follicular phase (FF) (2-7 days before egg pick-up), ovulatory phase (FO) (on the day of egg pick-up) and luteal phase (FL) (5-10 days after egg pick-up) in non-PCOS women undergoing ovarian stimulation and ICSI treatment (group 2).
Evaluation of the fluctuation of SP during the ovarian cycle in non-PCOS women undergoing ICSI treatment | 5 days before egg pick-up, day of egg pick up, 10 days after egg pick-up
  Assess the absolute difference of blood concentration of SP and the relative difference of its concentration [100 - (CFO*100/CFF) and 100 - (CFL*100/CFO)] in the three phases of the ovarian cycle: follicular phase (FF) (2-7 days before egg pick-up), ovulatory phase (FO) (on the day of egg pick-up) and luteal phase (FL) (5-10 days after egg pick-up) in non-PCOS women undergoing ovarian stimulation and ICSI treatment (group 2).
Evaluation of the fluctuation of enkephalins during the ovarian cycle in non-PCOS women undergoing ICSI treatment | 5 days before egg pick-up, day of egg pick up, 10 days after egg pick-up
  Assess the absolute difference of blood concentration of enkephalins and the relative difference of its concentration [100 - (CFO*100/CFF) and 100 - (CFL*100/CFO)] in the three phases of the ovarian cycle: follicular phase (FF) (2-7 days before egg pick-up), ovulatory phase (FO) (on the day of egg pick-up) and luteal phase (FL) (5-10 days after egg pick-up) in non-PCOS women undergoing ovarian stimulation and ICSI treatment (group 2).
Evaluation of the fluctuation of VIP during the ovarian cycle in non-PCOS women undergoing ICSI treatment | 5 days before egg pick-up, day of egg pick up, 10 days after egg pick-up
  Assess the absolute difference of blood concentration of VIP and the relative difference of its concentration [100 - (CFO*100/CFF) and 100 - (CFL*100/CFO)] in the three phases of the ovarian cycle: follicular phase (FF) (2-7 days before egg pick-up), ovulatory phase (FO) (on the day of egg pick-up) and luteal phase (FL) (5-10 days after egg pick-up) in non-PCOS women undergoing ovarian stimulation and ICSI treatment (group 2).
Evaluation of the fluctuation of CGRP during the ovarian cycle in PCOS women undergoing ICSI treatment | 5 days before egg pick-up, day of egg pick up, 10 days after egg pick-up
  Assess the absolute difference in blood concentration of CGRP and the relative difference in its concentration [100 - (CFO*100/CFF) and 100 - (CFL*100/CFO)] in the three phases of the ovarian cycle: follicular phase (FF) (2-7 days before oocyte pick-up), ovulatory phase (FO) (on the day of oocyte pick-up) and luteal phase (FL) (5-10 days after oocyte pick-up) in PCOS women undergoing ovarian stimulation procedure and ICSI treatment (group 3).
Evaluation of the fluctuation of SP during the ovarian cycle in PCOS women undergoing ICSI treatment | 5 days before egg pick-up, day of egg pick up, 10 days after egg pick-up
  Assess the absolute difference in blood concentrations of SP and the relative difference in its concentration [100 - (CFO*100/CFF) and 100 - (CFL*100/CFO)] in the three phases of the ovarian cycle: follicular phase (FF) (2-7 days before oocyte pick-up), ovulatory phase (FO) (on the day of oocyte pick-up) and luteal phase (FL) (5-10 days after oocyte pick-up) in PCOS women undergoing ovarian stimulation procedure and ICSI treatment (group 3).
Evaluation of the fluctuation of enkephalins during the ovarian cycle in PCOS women undergoing ICSI treatment | 5 days before egg pick-up, day of egg pick up, 10 days after egg pick-up
  Assess the absolute difference in blood concentration of enkephalins and the relative difference in its concentration [100 - (CFO*100/CFF) and 100 - (CFL*100/CFO)] in the three phases of the ovarian cycle: follicular phase (FF) (2-7 days before oocyte pick-up), ovulatory phase (FO) (on the day of oocyte pick-up) and luteal phase (FL) (5-10 days after oocyte pick-up) in PCOS women undergoing ovarian stimulation procedure and ICSI treatment (group 3).
Evaluation of the fluctuation of VIP during the ovarian cycle in PCOS women undergoing ICSI treatment | 5 days before egg pick-up, day of egg pick up, 10 days after egg pick-up
  Assess the absolute difference in blood concentration of VIP and the relative difference in its concentration [100 - (CFO*100/CFF) and 100 - (CFL*100/CFO)] in the three phases of the ovarian cycle: follicular phase (FF) (2-7 days before oocyte pick-up), ovulatory phase (FO) (on the day of oocyte pick-up) and luteal phase (FL) (5-10 days after oocyte pick-up) in PCOS women undergoing ovarian stimulation procedure and ICSI treatment (group 3).
Comparison of CGRP blood concentration between PCOS women and non-PCOS women undergoing ICSI treatment | 5 days before egg pick-up, day of egg pick up, 10 days after egg pick-up
  Comparison of absolute and relative blood concentration of CGRP in the three phases of the ovarian cycle between group 2 (non-PCOS women undergoing ICSI) and group 3 (PCOS women undergoing ICSI), to assess whether, with the same ovulatory condition and treatment, there is increased and significant expression of CGRP in PCOS women compared with non-PCOS women.
Comparison of SP blood concentration between PCOS women and non-PCOS women undergoing ICSI treatment | 5 days before egg pick-up, day of egg pick up, 10 days after egg pick-up
  Comparison of absolute and relative blood concentration of SP in the three phases of the ovarian cycle between group 2 (non-PCOS women undergoing ICSI) and group 3 (PCOS women undergoing ICSI), to assess whether, with the same ovulatory condition and treatment, there is increased and significant expression of SP in PCOS women compared with non-PCOS women.
Comparison of enkephalins blood concentration between PCOS women and non-PCOS women undergoing ICSI treatment | 5 days before egg pick-up, day of egg pick up, 10 days after egg pick-up
  Comparison of absolute and relative blood concentration of enkephalins in the three phases of the ovarian cycle between group 2 (non-PCOS women undergoing ICSI) and group 3 (PCOS women undergoing ICSI), to assess whether, with the same ovulatory condition and treatment, there is increased and significant expression of enkephalins in PCOS women compared with non-PCOS women.
Comparison of VIP blood concentration between PCOS women and non-PCOS women undergoing ICSI treatment | 5 days before egg pick-up, day of egg pick up, 10 days after egg pick-up
  Comparison of absolute and relative blood concentration of VIP in the three phases of the ovarian cycle between group 2 (non-PCOS women undergoing ICSI) and group 3 (PCOS women undergoing ICSI), to assess whether, with the same ovulatory condition and treatment, there is increased and significant expression of VIP in PCOS women compared with non-PCOS women.
Comparison of CGRP blood concentration between non-PCOS women with normal ovarian cycle and non-PCOS women undergoing ICSI treatment | 7 days after menstruation, 14 days after menstruation, 20 days after menstruation
  Comparison of absolute and relative blood concentrations of CGRP in the three phases of the ovarian cycle between group 1 (control) and group 2 (non-PCOS women undergoing ICSI tratment), to assess whether, ovarian stimulation represents a modifying factor of neuropeptide expression.
Comparison of SP blood concentration between non-PCOS women with normal ovarian cycle and non-PCOS women undergoing ICSI treatment | 7 days after menstruation, 14 days after menstruation, 20 days after menstruation
  Comparison of absolute and relative blood concentrations of SP in the three phases of the ovarian cycle between group 1 (control) and group 2 (non-PCOS women undergoing ICSI tratment), to assess whether, ovarian stimulation represents a modifying factor of neuropeptide expression.
Comparison of enkephalins blood concentration between non-PCOS women with normal ovarian cycle and non-PCOS women undergoing ICSI treatment | 7 days after menstruation, 14 days after menstruation, 20 days after menstruation
  Comparison of absolute and relative blood concentrations of enkephalins in the three phases of the ovarian cycle between group 1 (control) and group 2 (non-PCOS women undergoing ICSI tratment), to assess whether, ovarian stimulation represents a modifying factor of neuropeptide expression.
Comparison of VIP blood concentration between non-PCOS women with normal ovarian cycle and non-PCOS women undergoing ICSI treatment | 7 days after menstruation, 14 days after menstruation, 20 days after menstruation
  Comparison of absolute and relative blood concentrations of VIP in the three phases of the ovarian cycle between group 1 (control) and group 2 (non-PCOS women undergoing ICSI tratment), to assess whether, ovarian stimulation represents a modifying factor of neuropeptide expression.
Comparison of CGRP concentration in follicolar fluid between non-PCOS women and PCOS women both undergoing ICSI treatment | 5 days before egg pick-up, day of egg pick up, 10 days after egg pick-up
  Evaluate in PCOS and non-PCOS women undergoing ICSI tratment whether CGRP are released into the follicular fluid. If yes, compare absolute and relative concentrations of CGRP between the two groups and assess whether there is a correlation between oocyte quality and neuropeptide dosage.
Comparison of SP concentration in follicolar fluid between non-PCOS women and PCOS women both undergoing ICSI treatment | 5 days before egg pick-up, day of egg pick up, 10 days after egg pick-up
  Evaluate in PCOS and non-PCOS women undergoing ICSI tratment whether SP are released into the follicular fluid. If yes, compare absolute and relative concentrations of CGRP between the two groups and assess whether there is a correlation between oocyte quality and neuropeptide dosage.
Comparison of enkephalins concentration in follicolar fluid between non-PCOS women and PCOS women both undergoing ICSI treatment | 5 days before egg pick-up, day of egg pick up, 10 days after egg pick-up
  Evaluate in PCOS and non-PCOS women undergoing ICSI tratment whether enkephalins are released into the follicular fluid. If yes, compare absolute and relative concentrations of CGRP between the two groups and assess whether there is a correlation between oocyte quality and neuropeptide dosage.
Comparison of VIP concentration in follicolar fluid between non-PCOS women and PCOS women both undergoing ICSI treatment | 5 days before egg pick-up, day of egg pick up, 10 days after egg pick-up
  Evaluate in PCOS and non-PCOS women undergoing ICSI tratment whether VIP are released into the follicular fluid. If yes, compare absolute and relative concentrations of CGRP between the two groups and assess whether there is a correlation between oocyte quality and neuropeptide dosage.

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Gerli, Professor, Principal Investigator — University Of Perugia
Locations (1):
- University of Perugia, Piazza Menghini 1, S. Andrea delle Fratte., Perugia, Umbria, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] International evidence-based guidelines for the assessment and management of polycystic ovary syndrome 2018. Melbourne, Monash University
- [Background] Slowey MJ. Polycystic ovary syndrome: new perspective on an old problem. South Med J. 2001 Feb;94(2):190-6. PMID 11235033
- [Background] Pasquali R. Metabolic Syndrome in Polycystic Ovary Syndrome. Front Horm Res. 2018;49:114-130. doi: 10.1159/000485995. Epub 2018 Apr 5. PMID 29894990
- [Background] Tekin G, Tekin A, Kilicarslan EB, Haydardedeoglu B, Katircibasi T, Kocum T, Erol T, Colkesen Y, Sezgin AT, Muderrisoglu H. Altered autonomic neural control of the cardiovascular system in patients with polycystic ovary syndrome. Int J Cardiol. 2008 Oct 30;130(1):49-55. doi: 10.1016/j.ijcard.2007.08.037. Epub 2007 Dec 4. PMID 18055040
- [Background] Sverrisdottir YB, Mogren T, Kataoka J, Janson PO, Stener-Victorin E. Is polycystic ovary syndrome associated with high sympathetic nerve activity and size at birth? Am J Physiol Endocrinol Metab. 2008 Mar;294(3):E576-81. doi: 10.1152/ajpendo.00725.2007. Epub 2008 Jan 15. PMID 18198350
- [Background] Morales-Ledesma L, Trujillo Hernandez A, Ramirez MI, Rosas G, Linares R. Administration of a VIP-antagonist in vivo modifies ovarian hormone secretion in a rat model with polycystic ovary syndrome. Life Sci. 2021 Jan 15;265:118792. doi: 10.1016/j.lfs.2020.118792. Epub 2020 Nov 18. PMID 33220286
- [Background] Ilie IR. Neurotransmitter, neuropeptide and gut peptide profile in PCOS-pathways contributing to the pathophysiology, food intake and psychiatric manifestations of PCOS. Adv Clin Chem. 2020;96:85-135. doi: 10.1016/bs.acc.2019.11.004. Epub 2019 Dec 12. PMID 32362321
- [Background] Moore AM, Campbell RE. Polycystic ovary syndrome: Understanding the role of the brain. Front Neuroendocrinol. 2017 Jul;46:1-14. doi: 10.1016/j.yfrne.2017.05.002. Epub 2017 May 25. PMID 28551304
- [Background] Kozlowska A, Wojtkiewicz J, Majewski M, Jana B. Localization of substance P, calcitonin gene related peptide and galanin in the nerve fibers of porcine cystic ovaries. Folia Histochem Cytobiol. 2011;49(4):622-30. doi: 10.5603/fhc.2011.0085. PMID 22252756
- [Background] Zhang Z, Gong F, Lu GX. Plasma level of calcitonin gene-related peptide in patients with polycystic ovary syndrome and its relationship to hormonal and metabolic parameters. Peptides. 2012 Apr;34(2):343-8. doi: 10.1016/j.peptides.2012.01.018. Epub 2012 Jan 31. PMID 22314079